CLINICAL TRIAL: NCT03689972
Title: A Randomized, Controlled, Open-Label, Rater-Blinded, Phase 3b Study of the Efficacy, Safety, and Tolerability of 6-Week Extended Interval Dosing (EID) of Natalizumab (BG00002) in Subjects With Relapsing-Remitting Multiple Sclerosis Switching From Treatment With 4-Week Natalizumab Standard Interval Dosing (SID) in Relation to Continued SID Treatment - Followed by an Open-Label Crossover Extension Study Comprising Subcutaneous and Intravenous Natalizumab Administration
Brief Title: A Study to Evaluate Efficacy, Safety, and Tolerability of EID of Natalizumab (BG00002) in Participants With RRMS Switching From Treatment With Natalizumab SID in Relation to Continued SID Treatment- Followed by Extension Study Comprising SC and IV Natalizumab Administration
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Biogen (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 101MS329; 2018-002145-11 (EudraCT Number)
Record Dates: First submitted 2018-09-27; First posted 2018-10-01 (Actual); Results first posted 2024-06-12 (Actual); Last update posted 2024-06-12 (Actual); Status verified 2024-05

CONDITIONS: Multiple Sclerosis, Relapsing-Remitting
MeSH Terms: conditions — Multiple Sclerosis, Relapsing-Remitting | interventions — Natalizumab

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (5):
- Part 1: IV Q4W (Experimental): Participants received natalizumab 300 mg intravenous (IV) infusion once Q4W up to Week 72.
  Interventions: Drug: Natalizumab
- Part 1: IV Q6W (Experimental): Participants received natalizumab 300 mg IV infusion once Q6W up to Week 72.
  Interventions: Drug: Natalizumab
- Part 2: Run-in Period: IV Q6W (Experimental): Participants who completed Part 1 or were newly enrolled in Part 2 received natalizumab 300 mg IV infusion Q6W from Week 72 through Week 102.
  Interventions: Drug: Natalizumab
- Part 2: Crossover Period: IV Q6W, then SC Q6W (Experimental): Participants who completed run-in period of Part 2 were randomized to receive natalizumab 300 mg IV infusion Q6W from Week 108 through Week 126 followed by natalizumab 300 mg subcutaneous (SC) injection Q6W from Week 132 through Week 150 along with a single dose of natalizumab 300 mg SC injection or IV infusion as per participant's choice at Week 156.
  Interventions: Drug: Natalizumab
- Part 2: Crossover Period: SC Q6W, then IV Q6W (Experimental): Participants who completed run-in period of Part 2 were randomized to receive natalizumab 300 mg SC injection Q6W from Week 108 through Week 126 followed by natalizumab 300 mg IV infusion Q6W from Week 132 through Week 150 along with a single dose of natalizumab 300 mg SC injection or IV infusion as per participant's choice at Week 156.
  Interventions: Drug: Natalizumab

INTERVENTIONS:
Drug: Natalizumab — Natalizumab 300 mg IV infusion.
  Other Names: BG00002
  Arms: Part 1: IV Q4W; Part 1: IV Q6W; Part 2: Run-in Period: IV Q6W
Drug: Natalizumab — Natalizumab 300 mg SC injection or IV infusion.
  Other Names: BG00002
  Arms: Part 2: Crossover Period: IV Q6W, then SC Q6W; Part 2: Crossover Period: SC Q6W, then IV Q6W

SUMMARY:
Part 1: The primary objective is to evaluate the efficacy of natalizumab extended interval dosing (EID) (every 6 weeks [Q6W]) in participants who have previously been treated with natalizumab standard interval dosing (SID) (every 4 weeks [Q4W]) for at least 12 months, in relation to continued Q4W treatment. The secondary objectives is to evaluate relapse-based clinical efficacy measures, disability worsening, additional Magnetic resonance imaging (MRI)-lesion efficacy measures and safety of Q6W in participants who have previously been treated with natalizumab Q4W for at least 12 months, in relation to continued Q4W treatment.

Part 2: The primary objective is to evaluate participant preference for subcutaneous (SC) versus intravenous (IV) route of natalizumab administration. The secondary objectives is to evaluate treatment satisfaction, drug preparation and administration time, safety and immunogenicity, efficacy and characterize pharmacokinetic (PK) and pharmacodynamic (PD) drug preparation and administration time of SC versus IV routes of natalizumab administration.

DETAILED DESCRIPTION:
This study will be conducted in 2 parts. At the end of part 1, participants who provide consent and are eligible, and newly enrolled participants, will enter part 2, an Open Label Extension comprising a crossover analysis.

Those participants who completed part 1 and cannot participate, or elect not to participate, in Part 2 (Open label extension) will enter a 12-week follow-up.

ELIGIBILITY:
Key Inclusion Criteria:

For Part 1:

* Ability of the participant to understand the purpose and risks of the study and provide signed and dated informed consent and authorization to use confidential health information in accordance with national and local participant privacy regulations.
* Diagnosis of relapsing remitting multiple sclerosis (RRMS) according to the McDonald criteria [Thompson 2018].
* Treatment with natalizumab as disease-modifying monotherapy for RRMS that is consistent with the approved dosing for a minimum of 12 months prior to randomization. The participant must have received at least 11 doses of natalizumab in the 12 months prior to randomization with no missed doses in the 3 months prior to randomization.
* Expanded Disability Status Scale (EDSS) score <=5.5 at screening.
* No relapses in the last 12 months prior to randomization, as determined by the enrolling Investigator.

For Part 2:

* Ability of the participants to understand the purpose and risks of the study and provide signed and dated informed consent for Part 2 and authorization to use confidential health information in accordance with national and local participant privacy regulations.
* Completed Part 1 Week 72 visit while remaining on their randomized treatment assignment of Q4W or Q6W.

Key Exclusion Criteria:

For Part 1:

* Primary and secondary progressive multiple sclerosis (MS).
* MRI positive for Gd-enhancing lesions at screening.
* Participants for whom MRI is contraindicated (e.g., have a contraindicated pacemaker or other contraindicated implanted metal device, have suffered, or are at risk for, side effects from Gd, or have claustrophobia that cannot be medically managed).
* History of any clinically significant (as determined by the Investigator) cardiac, endocrinologic, hematologic, hepatic, immunologic, metabolic (including diabetes), urologic, pulmonary, neurologic (except for RRMS), dermatologic, psychiatric, renal, or other major disease that would preclude participation in a clinical study, in the opinion of the Investigator.
* Presence of anti-natalizumab antibodies at screening.

For Part 2:

* Participants treated with natalizumab Q6W was reverted to natalizumab Q4W by choice or as rescue treatment in Part 1.
* Participant received treatment with any MS disease-modifying therapy other than natalizumab in Part 1 or in the period between Part 1 and Part 2.
* History of human immunodeficiency virus or history of other immunodeficient conditions.
* Current enrollment or a plan to enroll in any interventional clinical study in which an investigational treatment or approved therapy for investigational use is administered within 30 days (or 5 half-lives of the agent, whichever is longer) prior to the Baseline Visit or at any time during this study.
* Inability to comply with study requirements.
* Other unspecified reasons that, in the opinion of the Investigator or Biogen, make the participant unsuitable for enrollment.

The inclusion and exclusion criteria for new participants who did not participate in Part 1 of the study are the same as those for participants who did participate in Part 1.

NOTE: Other protocol defined Inclusion/Exclusion criteria may apply

Ages: 18 Years to 60 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 585 (Actual)
Dates: Start 2018-11-27 (Actual); Primary Completion 2023-01-31 (Actual); Study Completion 2023-07-24 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Medical Director, Study Director — Biogen
Locations (107):
- United States (52):
  - North Central Neurology Associates, P.C., Cullman, Alabama
  - Alabama Neurology Associates, Homewood, Alabama
  - UCI MIND, Irvine, California
  - UC San Diego Movement Disorder Center, La Jolla, California
  - MS Center of California, Laguna Hills, California
  - Stanford Hospital and Clinics, Palo Alto, California
  - University of Colorado Hospital Anschutz Outpatient Pavillion, Aurora, Colorado
  - Advanced Neurosciences Research, Fort Collins, Colorado
  - Yale University, Fairfield, Connecticut
  - Georgetown University Hospital-Medstar, Washington D.C., District of Columbia
  - University of Miami Miller School of Medicine, Miami, Florida
  - Infinity Clinical Research, LLC, Sunrise, Florida
  - University of South Florida, Tampa, Florida
  - Shepherd Center, Inc., Atlanta, Georgia
  - Atlanta Neuroscience Institute, Atlanta, Georgia
  - NorthShore University HealthSystem, Evanston, Illinois
  - Northwestern University, Evanston, Illinois
  - College Park Family Care Center, Overland Park, Kansas
  - Lahey Clinic Inc. - PARENT ACCOUNT, Burlington, Massachusetts
  - Neurology Center of New England P.C., Foxborough, Massachusetts
  - Beth Israel Deaconess Medical Center, Inc., Jamaica Plain, Massachusetts
  - Dragonfly Research, LLC, Wellesley, Massachusetts
  - South Shore Neurology Associates, Weymouth, Massachusetts
  - Michigan Institute for Neurological Disorders, Farmington Hills, Michigan
  - Michigan State University, Grand Rapids, Michigan
  - Memorial Healthcare, Owosso, Michigan
  - Minneapolis Clinic of Neurology, Golden Valley, Minnesota
  - Washington University, School of Medicine, St Louis, Missouri
  - Cleveland Clinic Lou Ruvo Center for Brain Health, Las Vegas, Nevada
  - RWJ Barnabas Health, Newark, New Jersey
  - Holy Name Medical Center, Teaneck, New Jersey
  - NYU Langone Clinical Cancer Center, New York, New York
  - Mount Sinai Medical Center, New York, New York
  - Columbia University Hervert Irving Comprehensive Cancer Center, New York, New York
  - Island Neurological Associates, P.C., Plainview, New York
  - Raleigh Neurology Associates, Raleigh, North Carolina
  - Wake Forest University Health Sciences, Winston-Salem, North Carolina
  - University of Cincinnati, Cincinnati, Ohio
  - The Cleveland Clinic Foundation, Cleveland, Ohio
  - OhioHealth Riverside Methodist Hospital, Columbus, Ohio
  - Dayton Center for Neurological Disorders, Dayton, Ohio
  - Providence Neurological Specialties, Portland, Oregon
  - Thomas Jefferson University, Philadelphia, Pennsylvania
  - Magee-Womens Hospital of UPMC, Pittsburgh, Pennsylvania
  - Sibyl Wray, MD Neurology, PC, Knoxville, Tennessee
  - Vanderbilt University Medical Center, Nashville, Tennessee
  - Central Texas Neurology Consultants, Round Rock, Texas
  - Rocky Mountain MS Research Group LLC, Salt Lake City, Utah
  - University Of Virginia, Charlottesville, Virginia
  - Multiple Sclerosis Center of Greater Washington, Vienna, Virginia
  - Virginia Mason Medical Center, Seattle, Washington
  - Wheaton Franciscan Healthcare, Milwaukee, Wisconsin
- Australia (6):
  - Royal North Shore Hospital, St Leonards, New South Wales
  - Brain and Mind Centre, Sydney, New South Wales
  - Lyell McEwin Hospital, Elizabeth Vale, South Australia
  - Box Hill Hospital, Box Hill, Victoria
  - The Alfred Hospital, Melbourne, Victoria
  - Royal Melbourne Hospital, Parkville, Victoria
- Belgium (4):
  - Cliniques Universitaires de Bruxelles Hopital Erasme, Brussels
  - Cliniques Universitaires Saint-Luc, Brussels
  - UZA, Edegem
  - CHU de Tivoli, La Louvière
- Canada (5):
  - St. Michael's Hospital, Toronto, Ontario
  - Clinique Neuro-Outaouais, Gatineau, Quebec
  - Recherche SEPMUS, Greenfield Park, Quebec
  - CHUM Centre de Recherche, Montreal, Quebec
  - Montreal Neurological Institute Clinical Research Unit, Montreal, Quebec
- France (6):
  - Groupe Hospitalier Pellegrin - Hôpital Pellegrin, Bordeaux
  - CHU CAEN - Hôpital de la Côte de Nacre, Caen
  - Hopital Roger Salengro - CHU Lille, Lille
  - CHU Nice - Hôpital Pasteur, Nice
  - CHU Nantes - Hopital Nord Laënnec, Saint-Herblain
  - CHU Strasbourg - Nouvel Hôpital Civil, Strasbourg
- Germany (10):
  - Neurologie im Alphamed, Bamberg
  - Charité - Campus Charité Mitte, Berlin
  - Katholisches Klinikum Bochum gGmbH, Bochum
  - Neuro Centrum Science GmbH, Erbach im Odenwald
  - Universitaetsklinikum Essen, Essen
  - Universitaetsklinikum Freiburg, Freiburg im Breisgau
  - Universitaetsklinikum Giessen und Marburg GmbH Standort Marburg, Marburg
  - Klinikum rechts der Isar der TU Muenchen, Munich
  - Universitaetsklinikum Muenster, Münster
  - Synconcept GmbH - Neuro MVZ, Stuttgart
- Chaim Sheba Medical Center, Ramat Gan, Israel
- Italy (5):
  - Azienda Ospedaliero Universitaria Policlinico "Gaspare Rodolico - San Marco" (Presidio G. Rodolico), Catania
  - Fondazione Istituto G.Giglio di Cefalù, Cefalù
  - Fondazione IRCCS Istituto Neurologico Carlo Besta, Milan
  - Azienda Ospedaliera Universitaria- Università degli Studi della Campania "Luigi Vanvitelli", Napoli
  - I.R.C.C.S. Neuromed-Istituto Neurologico Mediterraneo, Pozzilli
- Netherlands (3):
  - Amphia Ziekenhuis, Molengracht, Breda
  - St. Antonius Ziekenhuis, Nieuwegein
  - Zuyderland Medisch Centrum - Sittard-Geleen, Sittard
- Spain (5):
  - Hospital Universitari Arnau de Vilanova, Lleida, Catalonia
  - Hospital Universitario Virgen de la Arrixaca, El Palmar, Murcia
  - Hospital Universitario Ramon y Cajal, Madrid
  - Hospital Regional Universitario de Malaga, Málaga
  - Hospital Universitario Virgen Macarena, Seville
- United Kingdom (10):
  - King's College Hospital, London, Greater London
  - The National Hospital for Neurology & Neurosurgery, London, Greater London
  - Walton Centre for Neurology & Neurosurgery., Liverpool, Merseyside
  - Queen Elizabeth University Hospital Campus, Glasgow, Strathclyde
  - Newcastle University- Clinical Ageing Research Unit, Newcastle upon Tyne, Tyne & Wear
  - Charing Cross Hospital, London
  - Nottingham University Hospital, Queen's Medical Centre, Nottingham
  - Salford Care Organisation, Salford
  - Royal Hallamshire Hospital, Sheffield
  - Morriston Hospital, Swansea

IPD SHARING:
Plan to Share IPD: No
Please refer data queries to DataSharing@biogen.com.

REFERENCES:
- [Derived] Foley JF, Defer G, Ryerson LZ, Cohen JA, Arnold DL, Butzkueven H, Cutter GR, Giovannoni G, Killestein J, Wiendl H, Li K, Dsilva L, Toukam M, Ferber K, Sohn J, Engelman H, Lasky T. Pharmacokinetics and Pharmacodynamics of Natalizumab 6-Week Dosing vs Continued 4-Week Dosing for Relapsing-Remitting Multiple Sclerosis. Neurol Neuroimmunol Neuroinflamm. 2024 Dec;11(6):e200321. doi: 10.1212/NXI.0000000000200321. Epub 2024 Oct 11. PMID 39393045
- [Derived] Wiendl H, Foley J, Defer G, Zhovtis Ryerson L, Cohen JA, Arnold DL, Butzkueven H, Cutter GR, Giovannoni G, Killestein J, Domingo-Horne R, Toukam M, Nunn A, Maghzi AH, Kuhelj R, Lasky T. Patient Preference for Subcutaneous Versus Intravenous Administration with Every-6-Week Natalizumab (Tysabri(R)) Dosing: NOVA Phase IIIb Extension Study (Part 2). Neurol Ther. 2024 Oct;13(5):1385-1401. doi: 10.1007/s40120-024-00647-0. Epub 2024 Jul 24. PMID 39046635
- [Derived] Foley JF, Defer G, Ryerson LZ, Cohen JA, Arnold DL, Butzkueven H, Cutter G, Giovannoni G, Killestein J, Wiendl H, Smirnakis K, Xiao S, Kong G, Kuhelj R, Campbell N; NOVA study investigators. Comparison of switching to 6-week dosing of natalizumab versus continuing with 4-week dosing in patients with relapsing-remitting multiple sclerosis (NOVA): a randomised, controlled, open-label, phase 3b trial. Lancet Neurol. 2022 Jul;21(7):608-619. doi: 10.1016/S1474-4422(22)00143-0. Epub 2022 Apr 25. PMID 35483387

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Participants were enrolled at the investigative sites in Australia, Belgium, Canada, France, Germany, Israel, Italy, Netherlands, Spain, the United Kingdom, and the United States from 27 November 2018 to 20 June 2021.
Pre-assignment Details: 585 participants were enrolled in the study, out of which 499 participants were randomized in Part 1. A total of 396 participants completed Part 1 of the study, out of which 67 participants entered Part 2 of the study. A total of 153 participants (including 86 new participants) entered Part 2 crossover period and 123 participants completed the study.
Groups:
- Part 1: Standard Interval Dosing (SID) (Every 4 Weeks [Q4W]) IV: Participants received natalizumab 300 mg intravenous (IV) infusion Q4W up to Week 72.
- Part 1: Extended Interval Dosing (EID) (Every 6 Weeks [Q6W]) IV: Participants received natalizumab 300 mg IV infusion Q6W up to Week 72.
- Part 2: Crossover Period: IV Q6W Then SC Q6W: Participants who completed run-in period of Part 2 were randomized to receive natalizumab 300 mg IV infusion Q6W from Week 108 through Week 126 followed by natalizumab 300 mg subcutaneous (SC) injection Q6W from Week 132 through Week 150 along with a single dose of natalizumab 300 mg SC injection or IV infusion as per participant's choice at Week 156.
- Part 2: Crossover Period: SC Q6W Then IV Q6W: Participants who completed run-in period of Part 2 were randomized to receive natalizumab 300 mg SC injection Q6W from Week 108 through Week 126 followed by natalizumab 300 mg IV infusion Q6W from Week 132 through Week 150 along with a single dose of natalizumab 300 mg SC injection or IV infusion as per participant's choice at Week 156.
Period: Part 1 (Day 1 up to Week 72)
Arm/Group | Part 1: Standard Interval Dosing (SID) (Every 4 Weeks [Q4W]) IV | Part 1: Extended Interval Dosing (EID) (Every 6 Weeks [Q6W]) IV | Part 2: Run-in Period: IV Q6W | Part 2: Crossover Period: IV Q6W Then SC Q6W | Part 2: Crossover Period: SC Q6W Then IV Q6W
Started | 248 | 251 | 0 | 0 | 0
Completed (Completed denotes the participants that completed the study treatment.) | 194 | 202 | 0 | 0 | 0
Not Completed | 54 | 49 | 0 | 0 | 0
Not completed — Adverse Event | 1 | 3 | 0 | 0 | 0
Not completed — Lost to Follow-up | 0 | 2 | 0 | 0 | 0
Not completed — Protocol-Defined Rescue Criteria | 0 | 6 | 0 | 0 | 0
Not completed — Developed Persistent Anti-Natalizumab Antibodies | 1 | 3 | 0 | 0 | 0
Not completed — Consent Withdrawn | 14 | 9 | 0 | 0 | 0
Not completed — Investigator Decision | 9 | 6 | 0 | 0 | 0
Not completed — Pregnancy | 5 | 1 | 0 | 0 | 0
Not completed — Unwilling to Comply With Protocol | 3 | 2 | 0 | 0 | 0
Not completed — Randomized but not Dosed | 1 | 1 | 0 | 0 | 0
Not completed — Reason not Specified | 20 | 16 | 0 | 0 | 0
Period: Part 2:Run-in Period (Week73uptoWeek107)
Arm/Group | Part 1: Standard Interval Dosing (SID) (Every 4 Weeks [Q4W]) IV | Part 1: Extended Interval Dosing (EID) (Every 6 Weeks [Q6W]) IV | Part 2: Run-in Period: IV Q6W | Part 2: Crossover Period: IV Q6W Then SC Q6W | Part 2: Crossover Period: SC Q6W Then IV Q6W
Started | 0 | 0 | 158 | 0 | 0
Completed | 0 | 0 | 153 | 0 | 0
Not Completed | 0 | 0 | 5 | 0 | 0
Not completed — Consent Withdrawn | 0 | 0 | 2 | 0 | 0
Not completed — Pregnancy | 0 | 0 | 1 | 0 | 0
Not completed — Reason not Specified | 0 | 0 | 2 | 0 | 0
Period: Part2CrossoverPeriod(Week108uptoWeek156)
Arm/Group | Part 1: Standard Interval Dosing (SID) (Every 4 Weeks [Q4W]) IV | Part 1: Extended Interval Dosing (EID) (Every 6 Weeks [Q6W]) IV | Part 2: Run-in Period: IV Q6W | Part 2: Crossover Period: IV Q6W Then SC Q6W | Part 2: Crossover Period: SC Q6W Then IV Q6W
Started | 0 | 0 | 0 | 75 | 78
Completed (Completed denotes the participants that completed the study treatment.) | 0 | 0 | 0 | 63 | 60
Not Completed | 0 | 0 | 0 | 12 | 18
Not completed — Adverse Event | 0 | 0 | 0 | 1 | 1
Not completed — Consent Withdrawn | 0 | 0 | 0 | 7 | 1
Not completed — Investigator Decision | 0 | 0 | 0 | 2 | 2
Not completed — Pregnancy | 0 | 0 | 0 | 0 | 1
Not completed — Reason not Specified | 0 | 0 | 0 | 2 | 1
Not completed — Randomized but not Dosed | 0 | 0 | 0 | 0 | 12

BASELINE CHARACTERISTICS:
Population: Part 1: All randomized population included all the randomized participants in Part 1 of the study. Part 2: Included all the newly enrolled randomized participants in the crossover period of Part 2 of the study.
Groups:
- Part 1: IV Q4W: Participants received natalizumab 300 mg IV infusion Q4W up to Week 72.
- Part 1: IV Q6W: Participants received natalizumab 300 mg IV infusion Q6W up to Week 72.
- Part 2: Crossover Period: Participants who were newly enrolled in Part 2 received natalizumab 300 mg IV infusion Q6W from Week 108 through Week 126 followed by natalizumab 300 mg SC injection Q6W from Week 132 through Week 150, or natalizumab 300 mg SC injection Q6W from Week 108 through Week 126 followed by natalizumab 300 mg IV infusion Q6W from Week 132 through Week 150, along with a single dose of natalizumab 300 mg SC injection or IV infusion as per participant's choice at Week 156.
- Total: Total of all reporting groups
Arm/Group | Part 1: IV Q4W | Part 1: IV Q6W | Part 2: Crossover Period | Total
Number analyzed (Participants) | 248 | 251 | 86 | 585
Age, Continuous [Mean (Standard Deviation); unit: Years] | 40.5 (10.03) | 41.0 (9.66) | 37.6 (9.85) | 40.3 (9.9)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 181 | 178 | 58 | 417
  Male | 67 | 73 | 28 | 168
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 10 | 9 | 1 | 20
  Not Hispanic or Latino | 223 | 224 | 67 | 514
  Unknown or Not Reported | 15 | 18 | 18 | 51
Race/Ethnicity, Customized [Count of Participants; unit: Participants]
  Race: American Indian or Alaska Native | 1 | 1 | 0 | 2
  Race: Asian | 1 | 4 | 0 | 5
  Race: Black or African American | 23 | 14 | 0 | 37
  Race: White | 211 | 211 | 71 | 493
  Race: Not Reported | 11 | 15 | 14 | 40
  Race: Other | 1 | 6 | 1 | 8

OUTCOME MEASURES:

1. Primary Outcome: Part 1: Mean Number of New or Newly Enlarging T2 Hyperintense Lesions at Week 72
Description: T2 hyperintense lesions were analyzed by magnetic resonance imaging (MRI) scans of brain. New MRI scans were compared with the prior MRI scans to analyze the number of new or newly enlarging T2 hyperintense lesions at Week 72 relative to baseline.
Time Frame: Week 72
Population: Modified intent to treat (mITT) population included all randomized participants who received at least one dose of study treatment and had at least one postbaseline result in Part 1. Here, 'overall number of participants analyzed' signifies the number of participants with data available for outcome measure analysis.
Measure: Mean (95% Confidence Interval); unit: number of T2 lesions
Arm/Group | Part 1: IV Q4W | Part 1: IV Q6W
Number analyzed (Participants) | 197 | 211
number of T2 lesions | 0.05 [0.01 to 0.22] | 0.20 [0.07 to 0.63]
Statistical Analysis 1: Comparison: Part 1: IV Q4W vs Part 1: IV Q6W; Test type: Superiority; p = 0.0755, Negative Binomial Regression; The model included treatment as classification variable & baseline body weight, duration of natalizumab exposure at baseline, & region as covariates; Ratio of Mean = 4.24, 95% CI 2-sided [0.86 to 20.85]

2. Primary Outcome: Part 2: Percentage of Participants Indicating a Preference for Natalizumab SC Administration at the End of Crossover Period of Part 2
Time Frame: Week 150
Population: mITT population included all randomized participants who received at least one dose of SC natalizumab after randomization in Part 2 and who completed at least the first question in the Patient Preference Questionnaire (PPQ) on one occasion. Here, 'overall number of participants analyzed' signifies the number of participants with data available for outcome measure analysis. (Confidence interval=CI)
Measure: Number; unit: percentage of participants
Groups:
- Part 2: Crossover Period: IV Q6W Then SC Q6W: Participants who completed run-in period of Part 2 were randomized to receive natalizumab 300 mg IV infusion Q6W from Week 108 through Week 126 followed by natalizumab 300 mg SC injection Q6W from Week 132 through Week 150 along with a single dose of natalizumab 300 mg SC injection or IV infusion as per participant's choice at Week 156.
Arm/Group | Part 2: Crossover Period: IV Q6W Then SC Q6W | Part 2: Crossover Period: SC Q6W Then IV Q6W
Number analyzed (Participants) | 62 | 61
percentage of participants | 83.9 | 91.8
Statistical Analysis 1: Comparison: Part 2: Crossover Period: IV Q6W Then SC Q6W vs Part 2: Crossover Period: SC Q6W Then IV Q6W; Test type: Superiority; Exact Binomial method; Percentage of participants preferring natalizumab SC at end of crossover period of Part 2, and 95% CI was calculated using the exact binomial method; Percentage = 87.8, 95% CI 2-sided [80.68 to 93.01]

3. Secondary Outcome: Part 1: Time to First Relapse as Adjudicated by an Independent Neurology Evaluation Committee (INEC)
Description: Relapse is defined as the onset of new or recurrent neurological symptoms, not associated with fever, infection, severe stress, or drug toxicity, lasting at least 24 hours, accompanied by new objective abnormalities on a neurological examination. Only relapses confirmed by an INEC were included in the analysis. Time to First Relapse was estimated by Kaplan-Meier method.
Time Frame: Up to Week 72
Population: mITT population included all randomized participants who received at least one dose of study treatment and had at least one postbaseline result in Part 1.
Measure: Median (Inter-Quartile Range); unit: weeks
Arm/Group | Part 1: IV Q4W | Part 1: IV Q6W
Number analyzed (Participants) | 242 | 247
weeks | NA [NA to NA] — Median, Q1 and Q3 were not reached in the Kaplan-Meier curve due to insufficient number of relapses. | NA [NA to NA] — Median, Q1 and Q3 were not reached in the Kaplan-Meier curve due to insufficient number of relapses.

4. Secondary Outcome: Part 1: Annualized Relapse Rate at Week 72
Description: Annualized relapse rate is calculated as the total number of INEC-confirmed relapses that occurred during the treatment period divided by the total number of participant-years followed in the period.
Time Frame: Week 72
Population: as for outcome 3
Measure: Number (95% Confidence Interval); unit: relapses per participant-year
Arm/Group | Part 1: IV Q4W | Part 1: IV Q6W
Number analyzed (Participants) | 242 | 247
relapses per participant-year | 0.00010 [0.00004 to 0.00024] | 0.0001 [0.00006 to 0.00027]
Statistical Analysis 1: Comparison: Part 1: IV Q4W vs Part 1: IV Q6W; Test type: Superiority; p = 0.6312, Poisson Regression; Poisson regression model was adjusted for baseline body weight, duration of natalizumab exposure at baseline, and region; Ratio of annualized relapse rate = 1.32481, 95% CI 2-sided [0.42016 to 4.17725]

5. Secondary Outcome: Part 1: Time to Expanded Disability Status Scale (EDSS) Worsening
Description: Confirmed EDSS worsening is defined as an increase of at least 1.0 point from a baseline EDSS score ≥ 1.0 or an increase of at least 1.5 points from a baseline EDSS score of 0 that is confirmed after at least 24 weeks. Time to EDSS worsening is estimated by Kaplan-Meier method.
Time Frame: Up to Week 72
Population: as for outcome 3
Measure: Median (Inter-Quartile Range); unit: weeks
Arm/Group | Part 1: IV Q4W | Part 1: IV Q6W
Number analyzed (Participants) | 242 | 247
weeks | NA [NA to NA] — Median, Q1, and Q3 were not reached in the Kaplan-Meier curve due to insufficient number of events. | NA [NA to NA] — Median, Q1, and Q3 were not reached in the Kaplan-Meier curve due to insufficient number of events.

6. Secondary Outcome: Part 1: Mean Number of New T1 Hypointense Lesions at Weeks 24, 48, and 72
Description: T1 hypointense lesions on brain were analyzed by MRI scans of brain. New MRI scans were compared with the prior MRI scans to analyze the number of new T1 hypointense lesions at Weeks 24, 48, and 72 relative to baseline.
Time Frame: Weeks 24, 48, and 72
Population: mITT population included all randomized participants who received at least one dose of study treatment and had at least one postbaseline result in Part 1. 'Overall number of participants analyzed' signifies the number of participants with data available for outcome measure analysis. Here, 'number analyzed' signifies the number of participants with data available for analysis at specified time-point.
Measure: Mean (Standard Deviation); unit: number of T1 lesions
Arm/Group | Part 1: IV Q4W | Part 1: IV Q6W
Number analyzed (Participants) | 227 | 241
number of T1 lesions
  Week 24 | 0.0 (0.13) | 0.0 (0.06)
  Week 48: number analyzed (Participants) | 202 | 218
  Week 48 | 0.0 (0.16) | 0.0 (0.07)
  Week 72: number analyzed (Participants) | 191 | 209
  Week 72 | 0.0 (0.16) | 0.0 (0.32)

7. Secondary Outcome: Part 1: Mean Number of New or Newly Enlarging T2 Hyperintense Lesions at Weeks 24 and 48
Description: T2 hyperintense lesions were analyzed by MRI scans of brain. New MRI scans were compared with the prior MRI scans to analyze the number of new or newly enlarging T2 hyperintense lesions at Weeks 24 and 48 relative to baseline.
Time Frame: Weeks 24 and 48
Population: mITT population included all randomized participants who received at least one dose of study treatment and had at least one postbaseline result in Part 1. 'Overall number of participants analyzed' signifies the number of participants with data available for outcome measure analysis. Here, 'number analyzed' signifies the number of participants with data available for analysis at specified time point.
Measure: Mean (Standard Deviation); unit: number of T2 lesions
Arm/Group | Part 1: IV Q4W | Part 1: IV Q6W
Number analyzed (Participants) | 229 | 242
number of T2 lesions
  Week 24 | 0.0 (0.16) | 0.0 (0.35)
  Week 48: number analyzed (Participants) | 206 | 221
  Week 48 | 0.0 (0.21) | 0.1 (1.03)

8. Secondary Outcome: Part 1: Mean Number of New Gadolinium (Gd) Enhancing Lesions at Weeks 24, 48, and 72
Description: Gd enhancing lesions on brain were analyzed by MRI scans of brain. New MRI scans were compared with the prior MRI scans to analyze the number of new Gd enhancing lesions at Weeks 24, 48, and 72 relative to baseline.
Time Frame: Weeks 24, 48, and 72
Population: as for outcome 6
Measure: Mean (Standard Deviation); unit: number of Gd lesions
Arm/Group | Part 1: IV Q4W | Part 1: IV Q6W
Number analyzed (Participants) | 227 | 241
number of Gd lesions
  Week 24 | 0.0 (0.07) | 0.0 (0.00)
  Week 48: number analyzed (Participants) | 203 | 218
  Week 48 | 0.0 (0.07) | 0.0 (0.00)
  Week 72: number analyzed (Participants) | 191 | 210
  Week 72 | 0.0 (0.07) | 0.1 (0.83)

9. Secondary Outcome: Part 1: Percentage of Participants With Treatment-Emergent Adverse Events (TEAEs) and Serious Adverse Events (SAEs)
Description: An AE is any untoward medical occurrence in a participant or clinical investigation participant administered a pharmaceutical product and that does not necessarily have a causal relationship with this treatment. An AE can therefore be any unfavorable and unintended sign (including an abnormal laboratory finding), symptom, or disease temporally associated with the use of a medicinal (investigational) product, whether or not related to the medicinal (investigational) product. A TEAE is any event occurring on or after first dose after randomization up to 12 weeks (or 24 weeks for PML [progressive multifocal leukoencephalopathy] events) following the last dose on the study.An SAE is any untoward medical occurrence that at any dose results in death, is a life-threatening event, requires inpatient hospitalization or prolongation of existing hospitalization, results in a significant disability/incapacity or congenital anomaly, is a medically important event.
Time Frame: Baseline up to Week 84
Population: Safety population included all randomized participants who received at least one dose of study treatment in Part 1.
Measure: Number; unit: percentage of participants
Arm/Group | Part 1: IV Q4W | Part 1: IV Q6W
Number analyzed (Participants) | 247 | 250
percentage of participants
  TEAEs | 76.9 | 77.6
  SAEs | 6.9 | 6.8

10. Secondary Outcome: Part 2: Change From Baseline in Treatment Satisfaction Questionnaire for Medication (TSQM) Scores During the Crossover Period
Description: The TSQM has 14 questions that assesses participants' global satisfaction level with their treatment in 4 domains: side effects (There are 5 questions in the side effects domain, however one of them is a Yes/No question and there are 4 sub-components, hence a maximum score of 20), effectiveness (3 questions), global satisfaction (3 questions), and convenience (3 questions). All questions are scored from 1 (least satisfied) to 5 or 7 (most satisfied). The total score is summed for each domain to obtain: side effects (1-20), effectiveness (1-21), global satisfaction (1-17), and convenience (1-21), using transformed scores between 0 and 100 for effectiveness. Lower total scores in each domain indicate dissatisfaction with the study medication and higher total scores indicate satisfaction.
Time Frame: Part 2 Baseline (Week 108) up to Week 156
Population: Full analysis set included all randomized participants who received at least one dose of study treatment during at least one study period and had at least one baseline assessment in Part 2. Here, 'overall number of participants analyzed' signifies the number of participants with data available for outcome measure analysis.
Measure: Least Squares Mean (Standard Error); unit: Score on a scale
Groups:
- Part 2: Crossover Period: IV Q6W: Participants received natalizumab 300 mg IV infusion Q6W for 24 weeks.
- Part 2: Crossover Period: SC Q6W: Participants received natalizumab 300 mg SC injection Q6W for 24 weeks.
Arm/Group | Part 2: Crossover Period: IV Q6W | Part 2: Crossover Period: SC Q6W
Number analyzed (Participants) | 127 | 127
Score on a scale | 0.17 (0.899) | 0.64 (0.902)
Statistical Analysis 1: Comparison: Part 2: Crossover Period: IV Q6W vs Part 2: Crossover Period: SC Q6W; Test type: Superiority; p = 0.764, Linear Mixed Effects Model — Performed with factors:route of administration,period,sequence,body weight,duration of natalizumab exposure,stratification factor,baseline TSQM score; Difference = 0.47, 95% CI 2-sided [-2.61 to 3.54]

11. Secondary Outcome: Part 2: Mean Time for Drug Preparation and Drug Administration During the Crossover Period
Time Frame: Week 108 up to Week 156
Population: Full analysis set included all randomized participants who received at least one dose of study treatment during at least one study period and had at least one baseline assessment in Part 2.
Measure: Mean (Standard Deviation); unit: minutes
Arm/Group | Part 2: Crossover Period: IV Q6W | Part 2: Crossover Period: SC Q6W
Number analyzed (Participants) | 136 | 132
minutes
  Drug Preparation Time | 4.9 (3.86) | 0 (0)
  Drug Administration Time | 62.6 (10.45) | 4.3 (5.11)

12. Secondary Outcome: Part 2: Percentage of Participants With Treatment-Emergent Adverse Events (TEAEs)
Description: An AE is any untoward medical occurrence in a participant or clinical investigation participant administered a pharmaceutical product and that does not necessarily have a causal relationship with this treatment. An AE can therefore be any unfavorable and unintended sign (including an abnormal laboratory finding), symptom, or disease temporally associated with the use of a medicinal (investigational) product, whether or not related to the medicinal (investigational) product. A TEAE is any event occurring on or after first dose after randomization up to and including 12 weeks (or 24 weeks for PML events) following the last dose on the study.
Time Frame: Part 2: Baseline (Week 108) up to Week 180
Population: Safety population included all randomized participants who received at least one dose of study treatment during the crossover period of Part 2.
Measure: Number; unit: percentage of participants
Arm/Group | Part 2: Crossover Period: IV Q6W | Part 2: Crossover Period: SC Q6W
Number analyzed (Participants) | 136 | 132
percentage of participants | 57.4 | 62.9

13. Secondary Outcome: Part 2: Percentage of Participants With Anti-Natalizumab Antibodies During the Crossover Period
Time Frame: Part 2 Baseline (Week 108) up to Week 156
Population: Immunogenicity population included all participants who received at least one dose of SC or IV natalizumab and had at least one assessment for anti-drug antibody during crossover period of Part 2.
Measure: Number; unit: percentage of participants
Arm/Group | Part 2: Crossover Period: IV Q6W | Part 2: Crossover Period: SC Q6W
Number analyzed (Participants) | 136 | 132
percentage of participants | 0 | 0

14. Secondary Outcome: Part 2: Mean Number of New or Newly Enlarging T2 Hyperintense Lesions During the Crossover Period
Description: T2 hyperintense lesions were analyzed by MRI scans of brain. New MRI scans were compared with the prior MRI scans to analyze the number of new or newly enlarging T2 hyperintense lesions during the crossover period of Part 2 relative to baseline.
Time Frame: Part 2 Baseline (Week 108) up to Week 156
Population: as for outcome 10
Measure: Mean (Standard Deviation); unit: number of T2 lesions
Arm/Group | Part 2: Crossover Period: IV Q6W | Part 2: Crossover Period: SC Q6W
Number analyzed (Participants) | 131 | 128
number of T2 lesions | 0.0 (0.09) | 0.0 (0.22)

15. Secondary Outcome: Part 2: Time to First Relapse During the Crossover Period
Description: Relapse is defined as the onset of new or recurrent neurological symptoms, not associated with fever, infection, severe stress, or drug toxicity, lasting at least 24 hours. The time to first relapse is defined as the time from the first randomized dose in Part 2 up to the first relapse. Time to First Relapse is estimated by Kaplan-Meier method.
Time Frame: Part 2 Baseline (Week 108) up to Week 156
Population: FAS: all randomized participants receiving ≥1 dose of study treatment during at least one study period and had ≥1 baseline assessment in Part 2. Overall number analyzed: participants without any relapse at beginning of crossover period of Part 2. As pre-specified in the Statistical Analysis Plan(SAP), time to event analyses was planned 'per treatment sequence' rather than 'per intervention' in Part 2 as protocol-specified analysis does not account for correlation of within participant effect.
Measure: Median (Inter-Quartile Range); unit: weeks
Arm/Group | Part 2: Crossover Period: IV Q6W Then SC Q6W | Part 2: Crossover Period: SC Q6W Then IV Q6W
Number analyzed (Participants) | 71 | 63
weeks | NA [NA to NA] — Median, Q1, and Q3 were not reached in the Kaplan-Meier curve due to one relapse. | NA [NA to NA] — Data is not available as no participant in this group had a relapse.

16. Secondary Outcome: Part 2: Annualized Relapse Rate During the Crossover Period
Description: Annualized relapse rate is calculated as the total number of relapses that occurred during the treatment period divided by the total number of participant-years followed in the period.
Time Frame: Part 2 Baseline (Week 108) up to Week 156
Population: Data was not analyzed for this outcome measure as only one relapse was observed in the Part 2 crossover period.
Arm/Group | Part 2: Crossover Period: IV Q6W Then SC Q6W | Part 2: Crossover Period: SC Q6W Then IV Q6W
Number analyzed (Participants) | 0 | 0

17. Secondary Outcome: Part 2: Change From Baseline in EDSS Score During the Crossover Period
Description: The EDSS is a scale based on standardized neurological examination which comprised of optic, brain stem, pyramidal, cerebellar, sensory and cerebral functions, as well as walking ability. It measures the MS disability status on a scale ranging from 0 (normal) to 10 (death due to MS), with higher scores indicating more disability.
Time Frame: Part 2 Baseline (Week 108) up to Week 156
Population: as for outcome 10
Measure: Least Squares Mean (Standard Error); unit: Score on a scale
Arm/Group | Part 2: Crossover Period: IV Q6W | Part 2: Crossover Period: SC Q6W
Number analyzed (Participants) | 135 | 132
Score on a scale | 0.02 (0.055) | 0.10 (0.056)
Statistical Analysis 1: Comparison: Part 2: Crossover Period: IV Q6W vs Part 2: Crossover Period: SC Q6W; Test type: Superiority; p = 0.357, Linear Mixed Effects Model — [p-value comment as in outcome 10, analysis 1]; Difference = 0.08, 95% CI 2-sided [-0.09 to 0.25]

18. Secondary Outcome: Part 2: Mean Number of New Gd Enhancing Lesions During the Crossover Period
Description: Gd enhancing lesions on brain were analyzed by MRI scans of brain. New MRI scans were compared with the prior MRI scans to analyze the number of new Gd enhancing lesions during the crossover period of Part 2 relative to baseline.
Time Frame: Week 108 up to Week 156
Population: as for outcome 10
Measure: Mean (Standard Deviation); unit: number of Gd lesions
Arm/Group | Part 2: Crossover Period: IV Q6W | Part 2: Crossover Period: SC Q6W
Number analyzed (Participants) | 131 | 128
number of Gd lesions | 0.0 (0.00) | 0.0 (0.00)

19. Secondary Outcome: Part 2: Mean Number of New T1 Hypointense Lesions During the Crossover Period
Description: T1 hypointense lesions on brain were analyzed by MRI scans of brain. New MRI scans were compared with the prior MRI scans to analyze the number of new T1 hypointense lesions during the crossover period of Part 2 relative to baseline.
Time Frame: Week 108 up to Week 156
Population: as for outcome 10
Measure: Mean (Standard Deviation); unit: number of T1 lesions
Arm/Group | Part 2: Crossover Period: IV Q6W | Part 2: Crossover Period: SC Q6W
Number analyzed (Participants) | 131 | 128
number of T1 lesions | 0.0 (0.09) | 0.0 (0.00)

20. Secondary Outcome: Part 2: Mean Percentage Change From Baseline in Brain Volume During the Crossover Period
Time Frame: Part 2 Baseline (Week 108) up to Week 156
Population: as for outcome 10
Measure: Least Squares Mean (Standard Error); unit: percent change
Arm/Group | Part 2: Crossover Period: IV Q6W | Part 2: Crossover Period: SC Q6W
Number analyzed (Participants) | 112 | 108
percent change | -0.11 (0.042) | -0.10 (0.042)

21. Secondary Outcome: Part 2: Change From Baseline in Cortical and Thalamic Brain Region Volume During the Crossover Period
Time Frame: Part 2 Baseline (Week 108) up to Week 156
Population: Full analysis set included all randomized participants who received at least one dose of study treatment during at least one study period and had at least one baseline assessment in Part 2. 'Overall number of participants analyzed' signifies the number of participants with data available for outcome measure analysis. Here "number analyzed" signifies the number of participants with data available for analysis at specified categories.
Measure: Least Squares Mean (Standard Error); unit: cubic centimeters (cm^3)
Arm/Group | Part 2: Crossover Period: IV Q6W | Part 2: Crossover Period: SC Q6W
Number analyzed (Participants) | 111 | 107
cubic centimeters (cm^3)
  Cortical Brain Region | -1478.82 (363.714) | -881.34 (367.155)
  Thalamic Brain Region: number analyzed (Participants) | 108 | 104
  Thalamic Brain Region | -25.98 (14.582) | -17.96 (14.796)

22. Secondary Outcome: Part 2: Trough Serum Concentration of Natalizumab (Ctrough) During the Crossover Period
Time Frame: Pre-dose at Weeks 108, 114, 120, 126, 132, 138, 144, 150, and 156
Population: Pharmacokinetic (PK) population included all participants who received at least one dose of SC or IV natalizumab and had at least one assessment for the concentration of natalizumab in serum during the crossover period of Part 2.
Measure: Mean (Standard Deviation); unit: micrograms per milliliter (µg/mL)
Arm/Group | Part 2: Crossover Period: IV Q6W | Part 2: Crossover Period: SC Q6W
Number analyzed (Participants) | 136 | 132
micrograms per milliliter (µg/mL) | 11.9 (11.50) | 10.3 (10.94)

23. Secondary Outcome: Part 2: Mean Trough α4 Integrin Saturation During the Crossover Period
Time Frame: Pre-dose at Weeks 108, 114, 120, 126, 132, 138, 144, 150, and 156
Population: Pharmacodynamic (PD) population included all participants who received at least one dose of SC or IV natalizumab after randomization in Part 2 and had at least one post-baseline assessment of the PD parameter. Here 'overall number of participants analyzed' indicates the number of participants without any relapse at the beginning of the crossover period of Part 2.
Measure: Mean (Standard Deviation); unit: percentage
Arm/Group | Part 2: Crossover Period: IV Q6W | Part 2: Crossover Period: SC Q6W
Number analyzed (Participants) | 135 | 132
percentage | 71.2 (15.31) | 67.2 (17.80)

ADVERSE EVENTS:
Time Frame: From first dose of study drug up to Week 180
Description: Safety population included all randomized participants who received at least one dose of study treatment. MedDRA version 24.0 applied for Part 1 and MedDRA version 26.0 applied for Part 2.
Arm/Group | Part 1: IV Q4W | Part 1: IV Q6W | Part 2: Run-in Period: IV Q6W | Part 2: Crossover Period: IV Q6W | Part 2: Crossover Period: SC Q6W
All-Cause Mortality (participants affected / at risk) | 0/247 | 0/250 | 0/158 | 0/136 | 0/132
Serious Adverse Events (participants affected / at risk) | 17/247 | 17/250 | 3/158 | 2/136 | 4/132
Other Adverse Events (participants affected / at risk) | 104/247 | 105/250 | 42/158 | 48/136 | 56/132
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Part 1: IV Q4W (N=247) | Part 1: IV Q6W (N=250) | Part 2: Run-in Period: IV Q6W (N=158) | Part 2: Crossover Period: IV Q6W (N=136) | Part 2: Crossover Period: SC Q6W (N=132)
Anaemia (Blood and lymphatic system disorders) | 1 | 0 | 0 | 0 | 0
Splenomegaly (Blood and lymphatic system disorders) | 0 | 0 | 1 | 0 | 0
Coronary artery dissection (Cardiac disorders) | 0 | 0 | 1 | 0 | 0
Goitre (Endocrine disorders) | 0 | 0 | 0 | 0 | 1
Papilloedema (Eye disorders) | 0 | 1 | 0 | 0 | 0
Diarrhoea (Gastrointestinal disorders) | 0 | 1 | 0 | 0 | 0
Hiatus hernia (Gastrointestinal disorders) | 0 | 0 | 0 | 1 | 0
Cholecystitis (Hepatobiliary disorders) | 0 | 1 | 0 | 0 | 0
Cholelithiasis (Hepatobiliary disorders) | 0 | 2 | 0 | 0 | 0
Drug hypersensitivity (Immune system disorders) | 1 | 0 | 0 | 0 | 0
Cholangitis infective (Infections and infestations) | 0 | 0 | 0 | 0 | 1
Covid-19 pneumonia (Infections and infestations) | 0 | 1 | 0 | 0 | 0
Gastroenteritis (Infections and infestations) | 1 | 0 | 0 | 0 | 0
Herpes zoster (Infections and infestations) | 1 | 0 | 0 | 0 | 0
Pneumonia (Infections and infestations) | 1 | 0 | 0 | 0 | 0
Progressive multifocal leukoencephalopathy (Infections and infestations) | 0 | 1 | 0 | 0 | 0
Respiratory tract infection (Infections and infestations) | 0 | 1 | 0 | 0 | 0
Ankle fracture (Injury, poisoning and procedural complications) | 0 | 1 | 0 | 0 | 0
Craniocerebral injury (Injury, poisoning and procedural complications) | 0 | 1 | 0 | 0 | 0
Fall (Injury, poisoning and procedural complications) | 1 | 1 | 0 | 0 | 0
Humerus fracture (Injury, poisoning and procedural complications) | 1 | 0 | 0 | 0 | 0
Post lumbar puncture syndrome (Injury, poisoning and procedural complications) | 1 | 0 | 0 | 0 | 0
Respiratory tract procedural complication (Injury, poisoning and procedural complications) | 0 | 1 | 0 | 0 | 0
Road traffic accident (Injury, poisoning and procedural complications) | 0 | 1 | 0 | 0 | 0
Tendon rupture (Injury, poisoning and procedural complications) | 0 | 1 | 0 | 0 | 0
Dehydration (Metabolism and nutrition disorders) | 0 | 1 | 0 | 0 | 0
Flank pain (Musculoskeletal and connective tissue disorders) | 0 | 1 | 0 | 0 | 0
Intervertebral disc protrusion (Musculoskeletal and connective tissue disorders) | 1 | 1 | 0 | 0 | 0
Osteoarthritis (Musculoskeletal and connective tissue disorders) | 1 | 0 | 0 | 0 | 0
Benign lung neoplasm (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0 | 0 | 0 | 0
Invasive ductal breast carcinoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 0 | 0 | 1 | 0
Leiomyoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0 | 0 | 0 | 0
Lipoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 1 | 0 | 0 | 0
Ovarian germ cell teratoma benign (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 0 | 0 | 0 | 1
Uterine leiomyoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0 | 0 | 0 | 0
Hemiparesis (Nervous system disorders) | 0 | 1 | 0 | 0 | 0
Lumbar radiculopathy (Nervous system disorders) | 1 | 0 | 0 | 0 | 0
Lumbosacral radiculopathy (Nervous system disorders) | 1 | 0 | 0 | 0 | 0
Migraine (Nervous system disorders) | 1 | 0 | 0 | 0 | 0
Multiple sclerosis pseudo relapse (Nervous system disorders) | 0 | 0 | 1 | 0 | 0
Multiple sclerosis relapse (Nervous system disorders) | 0 | 1 | 0 | 0 | 0
Neuropathy peripheral (Nervous system disorders) | 0 | 1 | 0 | 0 | 0
Optic neuritis (Nervous system disorders) | 0 | 0 | 1 | 0 | 0
Abortion (Pregnancy, puerperium and perinatal conditions) | 1 | 0 | 0 | 0 | 0
Depression (Psychiatric disorders) | 0 | 1 | 0 | 0 | 0
Suicidal ideation (Psychiatric disorders) | 0 | 1 | 0 | 0 | 0
Suicide attempt (Psychiatric disorders) | 0 | 1 | 0 | 0 | 0
Renal colic (Renal and urinary disorders) | 0 | 1 | 0 | 0 | 0
Ureterolithiasis (Renal and urinary disorders) | 1 | 0 | 0 | 0 | 0
Adnexal torsion (Reproductive system and breast disorders) | 0 | 0 | 0 | 0 | 1
Endometriosis (Reproductive system and breast disorders) | 1 | 0 | 0 | 0 | 0
Hyperventilation (Respiratory, thoracic and mediastinal disorders) | 1 | 0 | 0 | 0 | 0
Pneumothorax (Respiratory, thoracic and mediastinal disorders) | 0 | 1 | 0 | 0 | 0
Pulmonary embolism (Respiratory, thoracic and mediastinal disorders) | 1 | 0 | 0 | 0 | 0
Venous thrombosis limb (Vascular disorders) | 1 | 0 | 0 | 0 | 0
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | Part 1: IV Q4W (N=247) | Part 1: IV Q6W (N=250) | Part 2: Run-in Period: IV Q6W (N=158) | Part 2: Crossover Period: IV Q6W (N=136) | Part 2: Crossover Period: SC Q6W (N=132)
Fatigue (General disorders) | 8 | 25 | 4 | 3 | 2
Covid-19 (Infections and infestations) | 6 | 5 | 19 | 28 | 31
Nasopharyngitis (Infections and infestations) | 32 | 27 | 4 | 3 | 13
Upper respiratory tract infection (Infections and infestations) | 17 | 12 | 1 | 2 | 4
Urinary tract infection (Infections and infestations) | 19 | 24 | 6 | 7 | 2
Fall (Injury, poisoning and procedural complications) | 13 | 13 | 5 | 2 | 2
Arthralgia (Musculoskeletal and connective tissue disorders) | 9 | 18 | 1 | 2 | 8
Pain in extremity (Musculoskeletal and connective tissue disorders) | 7 | 14 | 4 | 1 | 1
Headache (Nervous system disorders) | 23 | 26 | 4 | 7 | 4
Cough (Respiratory, thoracic and mediastinal disorders) | 4 | 14 | 4 | 2 | 1

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
Our agreement is subject to confidentiality but generally the PI can publish, for non-commercial purposes only, results and methods of the trial, but no other Sponsor Confidential Information. PI must give Sponsor no less than 60 days to review any manuscript for a proposed publication and must delay publication for up to an additional 90 days thereafter if Sponsor needs to file any patent application to protect any of Sponsor's intellectual property contained in the proposed publication.

DOCUMENTS (2):
  • Study Protocol (2020-08-20): https://cdn.clinicaltrials.gov/large-docs/72/NCT03689972/Prot_000.pdf
  • Statistical Analysis Plan (2023-08-30): https://cdn.clinicaltrials.gov/large-docs/72/NCT03689972/SAP_001.pdf